CLINICAL TRIAL: NCT00785967
Title: Immune Responses to Neo-Antigens in Patients Treated With Raltegravir: Insights on V(D)J Recombination and RAG-1/2 Recombinase Function
Brief Title: Immune Responses in Patients Treated With Raltegravir
Acronym: RAG-1/2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unexpected and severe difficulties in recruitment.
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Chris Tsoukas, Director, Division of Allergy & CLinical Immunology, MUHC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MK0518-048-00, Version 2.2; HC-TPD Control # 120132
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: HIV Infections
Keywords: V(D)J recombination; RAG-1/2 recombinase function
MeSH Terms: conditions — HIV Infections | interventions — Hepatitis A Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine; E protein, bacteriophage X174

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): raltegravir 400mg bid + Truvada 1 tab qd
  Interventions: Biological: Various vaccines
- 2 (Active Comparator): efavirenz 600mg qhs + Truvada 1 tab qd (or Atripla 1 tab qhs)
  Interventions: Biological: Various vaccines

INTERVENTIONS:
Biological: Various vaccines — VAQTA: 1.0ml IM at weeks 24 & 48; Pneumovax 23: 0.5ml IM at screening; Td ADSORBED: 0.5ml IM at screening; phiX174 bacteriophage: 0.02ml/kg body weight IV at weeks 28, 32, 36, 40.
  Other Names: VAQTA;; Pneumovax 23;; Td ADSORBED;; phiX174 bacteriophage

SUMMARY:
Hypothesis: Treatment with raltegravir does not alter V(D)J recombination or immune responses to neoantigens.

A process known as V(D)J recombination is essential for developing lymphocytes and the specific functioning of the immune system. Raltegravir is the first approved drug of the new integrase inhibitor class of anti-HIV drugs. Integrase inhibitors have been shown in some studies to interfere with DNA cleavage and the activities of RAG-1/2. These studies suggest a potential to affect aspects of both B-cell and T-cell development, therefore, it is important to evaluate the potential effects that integrase inhibitors may have in clinical use. If immunoglobulin and T-cell receptor genes are altered by HIV integrase, then patient lymphocytes will fail to display normal responses to vaccinations.

DETAILED DESCRIPTION:
V(D)J recombination is essential for developing lymphocytes and the specific functioning of the immune system. Germline gene coding segments become rearranged to create functional immunoglobulin and T-cell receptor genes by this recombination. The process depends on site-specific cleavage of chromosomal DNA by RAG-1 and RAG-2 recombinase. Two recombination-activating gene proteins (RAG-1/2) in conjunction make up a complex of enzymes that join gene segments of B-cell and T-cell receptor genes. RAG-1 contains most of the V(D)J recombinase active site and RAG-2 is essential in joining DNA segments during V(D)J recombination. RAG-1/2 have similarity in action to other DNA transposases and HIV-1 integrase. These similarities suggest that HIV-1 integrase inhibitors may have the potential to affect aspects of both B-cell and T-cell development.

Induction of primary immune responses to neoantigens involves the generation of specific T-cells and immunoglobulin M (IgM) antibody secreting B-cells. As part of this process, T and B memory cells are also generated, which have specific cell surface receptors to the antigen. On repeat exposure to the antigen, these memory T- and B-cells are triggered to generate rapid and intense secondary responses. During this secondary response, B-cells secrete abundant specific IgG antibodies with greater affinity to the antigen than for the IgM isotope. This memory response is mediated by T-cells with CD45+ RO+ phenotype. These T-cells provide B-cells the help required to generate the specific IgG. Sub-optimal antibody responses are seen in both acquired and hereditary immunodeficiency, which are due to impaired T-cell function including poor T-helper responses to B-cells and defective neo-antigen responses.

An established method to evaluate T-cell function involves testing antibody production to vaccination with phiX174, a stable bacteriophage of E. Coli that is critical in demonstrating T-cell competence. Antibody titers after primary and secondary immunization correlate with abnormal CD4 cell help. Patients with functional B-cells that lack T-cell help show a characteristic failure to switch from IgM to IgG, making this assay essential in the evaluation of V(D)J recombination.

Currently, raltegravir is the only approved integrase inhibitor that targets the integration stage of the HIV-1 lifecycle. The clinical manifestations of raltegravir-related potential adverse effects on V(D)J recombination may be so rare that they may only be observed after large numbers of patients are exposed to this drug. Evaluating the direct in vivo interaction of HIV integrase inhibitors on RAG-1/2 is difficult, therefore the best approach may be to evaluate the potential negative effects on recombinase activity downstream by studying immune function. If gene rearrangements of immunoglobulin and T-cell receptor genes are altered by HIV integrase, then patient lymphocytes will fail to display normal responses to neo-antigen exposure. Since untreated HIV-infected individuals have an impaired ability to respond to new antigens, it is difficult to evaluate the responses to neo-antigens in these individuals. Therefore, to test this hypothesis, it would be best to choose patients with long-term control of HIV that have recovered immune function.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected males, as determined by ELISA and Western blot;
2. >18 years of age;
3. Current ARV therapy with efavirenz + Truvada® for >52 weeks;
4. HIV-1 RNA (bDNA) <50 copies/ml for at least 52 weeks;
5. No history of hepatitis A vaccine, and HAV antibody negative.

Exclusion Criteria:

1. any immunomodulatory therapy within 24 weeks of screening or during the trial;
2. any type of vaccine within 24 weeks of screening or during the trial;
3. current opportunistic infection, malignancy, acute infection, or febrile illness;
4. history of hypersensitivity to a vaccine, components of a vaccine, or components of a vaccine container.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Percent of patients with phiX174 IgG greater than or equal to 30% of total anti-phiX174 titers | Two weeks after fourth phiX174 immunization

SECONDARY OUTCOMES:
Total phiX174 antibody titers | 2 and 4 weeks after each immunization

CONTACTS AND LOCATIONS:
Overall Officials: Christos M Tsoukas, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Immune Deficiency Treatment Centre, Montreal General Hospital, McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Background] Melek M, Jones JM, O'Dea MH, Pais G, Burke TR Jr, Pommier Y, Neamati N, Gellert M. Effect of HIV integrase inhibitors on the RAG1/2 recombinase. Proc Natl Acad Sci U S A. 2002 Jan 8;99(1):134-7. doi: 10.1073/pnas.012610699. Epub 2001 Dec 26. PMID 11756686